CLINICAL TRIAL: NCT04394507
Title: Lymphatic Function and Interstitial Fluid Filtration in Patients With a Fontan Circulation From Brazil
Brief Title: Lymphatic Function in Patients With a Fontan Circulation From Brazil
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: InCor Heart Institute (Other); Hospital das Clínicas de Ribeirão Preto (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: Fontan Brazil
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Univentricular Heart; Lymphatic Abnormalities; Lymphatic Edema
Keywords: Lymphatic dysfunction; Near-Infrared Fluorescence Imaging; Fontan Circulation; Plethysmography
MeSH Terms: conditions — Univentricular Heart; Lymphatic Abnormalities; Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fontan Patients: Fontan patients operated at the two centres between 1991 and 2014.
  Interventions: Diagnostic Test: Near-Infrared Fluorescence imaging; Diagnostic Test: Strain Gauge Plethysmography
- Control Group: Age, gender and weight matched healthy controls.
  Interventions: Diagnostic Test: Near-Infrared Fluorescence imaging; Diagnostic Test: Strain Gauge Plethysmography

INTERVENTIONS:
Diagnostic Test: Near-Infrared Fluorescence imaging — .Near-infrared imaging was used to evaluate the function of the superficial lymphatic vessels in the right lower leg and foot as previously described.doi: 10.1161/CIRCIMAGING.118.008074.
Diagnostic Test: Strain Gauge Plethysmography — Strain Gauge Plethysmography to asses capillary filtration rate og the lower limb

SUMMARY:
It is suggested that the elevated central venous pressure in patients with a Fontan circulation can provoke manifestation of lymphatic dysfunction, met as plastic bronchitis, peripheral oedema and most feared protein-losing enteropathy (PLE).

An explorative study from our department at Aarhus University Hospital revealed that the function of the lymphatic vasculature in 10 young Fontan patients with no complications was abnormal compared to healthy controls. However, to further describe and confirm these findings we had to investigate the lymphatic circulation in a larger, older and more complicated group of Fontan patients.

The hypothesis is that, patients with a univentricular circulation have a reduced functionality of the lymphatic vasculature and which predisposes them to developing complications such as edema and PLE.

DETAILED DESCRIPTION:
The study population is patients with a Fontan circulation followed at InCor Heart Institute in Sao Paolo and Ribeirão Preto, Brazil. These were matched with and group of healthy controls.

The functional state of superficial lymphatics in the lower leg will be investigated, using near infrared fluorescence (NIRF) imaging. The capillary filtration of fluid and leakiness of the capillaries will be measured using strain gauge plethysmography and the peripheral blood flow will be measured using venous occlusion plethysmography. Furthermore, plasma concentration of noradrenaline will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Fontan circulation
* Age above 16.

Exclusion Criteria:

* Mental illness
* Syndromes.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients born with a univentricular heart treated surgically with a Fontan circulation in early childhood.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Lymphatic function assessed by Near-Infrared fluorescence Imaging 1 | 1 hour
  Contraction frequency (contraction/minut)
Lymphatic function assessed by Near-Infrared fluorescence Imaging 2 | 1 hour
  Pumping Pressure (mmHg)
Lymphatic function assessed by Near-Infrared fluorescence Imaging 3 | 1 hour
  Packet Velocity

SECONDARY OUTCOMES:
Capillary Filtration Rate measured by Strain Gauge Plethysmography | 1 hour
  Capillary Filtration Rate

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Hjortdal, MD, PhD, Dmsc, Study Director — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N, Central Jutland
  - Aarhus University, Aarhus C, Danmark

IPD SHARING:
Plan to Share IPD: No